CLINICAL TRIAL: NCT04625400
Title: Role of Bronchoscopy in Assessment of Patients With Post-intubation Tracheal Stenosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Darwish, Specialist , chest department and tuberculosis, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Tracheal stenosis
Record Dates: First submitted 2020-10-09; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Tracheal Stenosis
MeSH Terms: conditions — Tracheal Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- post intubation tracheal stenosis patients (Experimental): all ICU patients who were mechanically ventilated will be assessed for the possibility of presence of tracheal stenosis using spirometery and dyspnea will be assessed using (mMRC) score, chest X-ray to assess the location of tracheal stenosis and finally flexible bronchoscopy to confirm the presence of stenosis and identify the proper management.
  Interventions: Diagnostic Test: bronchoscope

INTERVENTIONS:
Diagnostic Test: bronchoscope — Bronchoscopy in Assessment of Patients With Post-intubation Tracheal Stenosis.

SUMMARY:
1. To estimate the importance of bronchoscopic treatment of tracheal stenosis and its effectiveness and safety.
2. To diagnose and evaluate tracheal stenosis characteristics as location, vertical extension and severity of obstruction.

DETAILED DESCRIPTION:
Post intubation tracheal stenosis (PI) was recognized in 1880, after prolonged endotracheal intubation in 4 patients with upper airway obstruction.The most common causes of acquired tracheal stenosis are endotracheal intubation and tracheostomy. Tracheal stenosis is a surgical problem managed non operatively by bronchoscopic dilation, endoluminal treatment with lasers, and stenting. Bronchoscopic management have a good success rate. PI and post tracheostomy stenosis (PT) are recognized with an 4.9 cases per million per year in the general population. Prolonged intubation can result in tracheal stenosis at various levels within the trachea.Tracheal stenosis occurs at the endotracheal tube cuff site in one third of the reported PI cases [9] and appears as a web-like fibrous. The mainly postulated cause is loss of regional blood flow.This injury begins within the first hours of intubation, and healing of the damaged areas within 3 to 6 weeks. Large volume, low pressure cuffs has reduced the occurrence of cuff injury.Patients in the ICU are common to have respiratory involvement, with 30-50% of the admissions requiring the use of mechanical ventilation.Flexible bronchoscopy has become the procedure of choice in most examinations of the tracheobronchial tree.The incidence of PI tracheal stenosis ranges from 6-21% and following tracheostomy ranges from 0.6-21%.

ELIGIBILITY:
Inclusion Criteria:

1. Meticulous History and Clinical Examination
2. Chest x-Ray (CXR)
3. Spirometry
4. Flexible bronchoscopy
5. Rigid Bronchoscopy (when needed).

Exclusion Criteria:

1. Patient refusal.
2. Any coagulation disorder.
3. Untreatable life-threatening arrhythmias.
4. Allergy to anaesthesia.
5. Poor general condition.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2021-01-01 (Estimated); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
tracheal stenosis incidence in ICU cases after mechanical ventilation | 2 years
  incidence of tracheal stenosis among ICU cases after mechanical ventilation assessed by flexible bronchoscope measured by numbers.(patients/year)

SECONDARY OUTCOMES:
the location, degree of tracheal stenosis characteristics. | 2 years
  1. identify the location of stenosis: - upper-third of the trachea (I) from 1-4 cm middle-third of the trachea (II) from 5-8 cm lower-third of the trachea (III)from 9-12 cm by Chest x-Ray (Chest x-ray)
  2. the diameter of trachea was assessed by cm.
  3. Spirometry by measuring the ratio of forced expiratory volume (FEV 1 ) in 1 second to peak expiratory flow (PEF).
  4. FEV 1 measured in in milliliter ,FEV1/FVC ratio.

CONTACTS AND LOCATIONS:
Overall Officials: Rafaat T El-Sokry, professor, Study Director — assuit university hospital

REFERENCES:
- [Result] Puchalski J, Musani AI. Tracheobronchial stenosis: causes and advances in management. Clin Chest Med. 2013 Sep;34(3):557-67. doi: 10.1016/j.ccm.2013.05.002. Epub 2013 Jul 3. PMID 23993823
- [Result] Galluccio G, Lucantoni G, Battistoni P, Paone G, Batzella S, Lucifora V, Dello Iacono R. Interventional endoscopy in the management of benign tracheal stenoses: definitive treatment at long-term follow-up. Eur J Cardiothorac Surg. 2009 Mar;35(3):429-33; discussion 933-4. doi: 10.1016/j.ejcts.2008.10.041. Epub 2008 Dec 11. PMID 19084420
- [Result] Cavaliere S, Bezzi M, Toninelli C, Foccoli P. Management of post-intubation tracheal stenoses using the endoscopic approach. Monaldi Arch Chest Dis. 2007 Jun;67(2):73-80. doi: 10.4081/monaldi.2007.492. PMID 17695689
- [Result] Mehta AC, Harris RJ, De Boer GE. Endoscopic management of benign airway stenosis. Clin Chest Med. 1995 Sep;16(3):401-13. PMID 8521696
- [Result] Mehta AC, Lee FY, Cordasco EM, Kirby T, Eliachar I, De Boer G. Concentric tracheal and subglottic stenosis. Management using the Nd-YAG laser for mucosal sparing followed by gentle dilatation. Chest. 1993 Sep;104(3):673-7. doi: 10.1378/chest.104.3.673. PMID 8365273
- [Result] Nouraei SA, Ma E, Patel A, Howard DJ, Sandhu GS. Estimating the population incidence of adult post-intubation laryngotracheal stenosis. Clin Otolaryngol. 2007 Oct;32(5):411-2. doi: 10.1111/j.1749-4486.2007.01484.x. No abstract available. PMID 17883582
- [Result] Poetker DM, Ettema SL, Blumin JH, Toohill RJ, Merati AL. Association of airway abnormalities and risk factors in 37 subglottic stenosis patients. Otolaryngol Head Neck Surg. 2006 Sep;135(3):434-7. doi: 10.1016/j.otohns.2006.04.013. PMID 16949978
- [Result] Pearson FG, Andrews MJ. Detection and management of tracheal stenosis following cuffed tube tracheostomy. Ann Thorac Surg. 1971 Oct;12(4):359-74. doi: 10.1016/s0003-4975(10)65137-5. No abstract available. PMID 4939117
- [Result] Grillo HC, Donahue DM, Mathisen DJ, Wain JC, Wright CD. Postintubation tracheal stenosis. Treatment and results. J Thorac Cardiovasc Surg. 1995 Mar;109(3):486-92; discussion 492-3. doi: 10.1016/S0022-5223(95)70279-2. PMID 7877309
- [Result] Weymuller EA Jr. Laryngeal injury from prolonged endotracheal intubation. Laryngoscope. 1988 Aug;98(8 Pt 2 Suppl 45):1-15. doi: 10.1288/00005537-198808001-00001. PMID 3398673
- [Result] Wain JC. Postintubation tracheal stenosis. Chest Surg Clin N Am. 2003 May;13(2):231-46. doi: 10.1016/s1052-3359(03)00034-6. PMID 12755310
- [Result] Ciccone AM, De Giacomo T, Venuta F, Ibrahim M, Diso D, Coloni GF, Rendina EA. Operative and non-operative treatment of benign subglottic laryngotracheal stenosis. Eur J Cardiothorac Surg. 2004 Oct;26(4):818-22. doi: 10.1016/j.ejcts.2004.06.020. PMID 15450579
- [Result] Estella A. Bronchoalveolar lavage for pandemic influenza A (H1N1)v pneumonia in critically ill patients. Intensive Care Med. 2010 Nov;36(11):1976-7. doi: 10.1007/s00134-010-2009-z. Epub 2010 Aug 6. No abstract available. PMID 20689914
- [Result] Anand VK, Alemar G, Warren ET. Surgical considerations in tracheal stenosis. Laryngoscope. 1992 Mar;102(3):237-43. doi: 10.1288/00005537-199203000-00002. PMID 1545649
- [Result] Grillo HC, Cooper JD, Geffin B, Pontoppidan H. A low-pressure cuff for tracheostomy tubes to minimize tracheal injury. A comparative clinical trial. J Thorac Cardiovasc Surg. 1971 Dec;62(6):898-907. No abstract available. PMID 4942973